CLINICAL TRIAL: NCT02642640
Title: Interaction of Melatonin and MTNR1B Genotype on Glucose Control - Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Frank AJL Scheer, PhD, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2015P000857A; R01DK102696 (NIH)
Record Dates: First submitted 2015-12-21; First posted 2015-12-30 (Estimated); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Glucose; Circadian Rhythm; Melatonin; Genes
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- melatonin-placebo (Other): subjects will receive melatonin first and placebo second
  Interventions: Dietary Supplement: melatonin; Drug: placebo
- placebo-melatonin (Other): subjects will receive placebo first and melatonin second
  Interventions: Dietary Supplement: melatonin; Drug: placebo

INTERVENTIONS:
Dietary Supplement: melatonin — 5 mg of melatonin per os.
Drug: placebo

SUMMARY:
This project aims to test the impact of melatonin and MTNR1B variation on regulation glucose regulation in a highly controlled in-laboratory setting and ex vivo in pancreatic islets.

DETAILED DESCRIPTION:
The investigators' recent GWAS discovery of MTNR1B as a novel type 2 diabetes gene has sparked great interest into the role of melatonin in glycemic control, for which the mechanism is largely unknown. This research will determine the effect of melatonin and MTNR1B on glycemic control under highly-controlled, in-laboratory protocols while manipulating circulating melatonin concentrations (both up and down) and assessing glycemic control by frequently-sampled intravenous glucose tolerance tests, as well as in ex vivo human pancreatic islets. This research will provide mechanistic insights into the metabolic effects of melatonin and the MTNR1B risk variant and may help in evidence-based approaches and personalized recommendations to improve glycemic control in night shift workers and late-night eaters.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index: 20 and 35 kg/m2
* Age: 21-55 years of age
* Caucasian
* Non-smoking
* With regular sleep-wake cycle
* Passed medical and psychological screening tests

Exclusion Criteria:

* Acute, chronic or debilitating medical conditions
* History of neurological or psychiatric disorder
* History of sleep disorder or regular use of sleep-promoting medication
* Current prescription, herbal, or over-the-counter medication use
* Traveling across 2 or more time zones within past 3 months
* Worked night or rotating shift work within past 1 year
* Drug or alcohol dependency

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-11; Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank AJL Scheer, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ambulatory phase (2/3 weeks), in which participants follow a self-selected Sleep-Wake cycle as well as eat pre-prepared, standardized meals for 3 days leading into the 5-day in-lab stay.
Period: Pre-in-lab phase
Arm/Group | Placebo-melatonin | Melatonin-placebo
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: Intervention 1
Arm/Group | Placebo-melatonin | Melatonin-placebo
Started | 12 | 11
Completed | 11 | 11
Not Completed | 1 | 0
Period: Washout
Arm/Group | Placebo-melatonin | Melatonin-placebo
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Intervention 2
Arm/Group | Placebo-melatonin | Melatonin-placebo
Started | 11 | 11
Completed | 11 | 10
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: baseline characteristics only used participants who completed the study
Groups:
- All Study Participants: All participants were randomized to receive all interventions, so all participants are combined into one Group "All Study Participants".
Arm/Group | All Study Participants
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
HbA1c [Mean (Standard Deviation); unit: %] | 5.2 (0.28)

OUTCOME MEASURES:

1. Primary Outcome: Disposition Index
Description: Disposition index is determined by frequently sampled intravenous glucose tolerance test. It is a composite measure of β-cell function adjusted for insulin sensitivity-was calculated as the product of insulin sensitivity and insulin secretion indices. High value means stronger β-cell function. Theoretical minimum is 0, no theoretical maximum.
Time Frame: During frequently sampled intravenous glucose tolerance test after melatonin/placebo administration on Day 2/4 (melatonin/placebo order randomized) in the laboratory visit
Population: 1 participant excluded at melatonin treatment because of a technical difficulty during one of the frequently sampled intravenous glucose tolerance tests
Measure: Geometric Mean (95% Confidence Interval); unit: index
Groups:
- Placebo: Placebo oral administration
- Melatonin: Melatonin oral administration
Arm/Group | Placebo | Melatonin
Number analyzed (Participants) | 21 | 20
index | 1314.7 [1012.6 to 1707.0] | 984.5 [687.0 to 1410.8]

2. Secondary Outcome: First-phase Beta-cell Responsivity
Description: First-phase beta-cell responsivity to glucose is determined by frequently sampled intravenous glucose tolerance test. It likely represents exocytosis of previously primed and docked insulin secretory granules (commonly called the readily releasable pool). It is given by the ratio between the incremental amount of C-peptide secreted during the first phase and the maximum increment of the plasma glucose concentration.High value means stronger β-cell responsivity. Theoretical minimum is 0, no theoretical maximum.
Time Frame: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: index
Arm/Group | Placebo | Melatonin
Number analyzed (Participants) | 21 | 21
index | 118.3 [98.3 to 142.4] | 88.9 [75.4 to 104.9]

3. Secondary Outcome: Insulin Sensitivity
Description: Insulin sensitivity is determined by frequently sampled intravenous glucose tolerance test. It is defined in quantitative terms as the effect of insulin to catalyse the disappearance of glucose from plasma.High value indicates better insulin sensitivity. Theoretical minimum is 0, no theoretical maximum.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: [(mu/l)^-1.min^-1]
Arm/Group | Placebo | Melatonin
Number analyzed (Participants) | 21 | 20
[(mu/l)^-1.min^-1] | 4.7 [3.7 to 5.8] | 3.7 [2.5 to 5.3]

4. Secondary Outcome: Glucose Tolerance
Description: glucose 3-hour incremental AUC during frequently sampled intravenous glucose tolerance test. High value indicates higher glucose level during the test, which is bad. Theoretical minimum is 0, no theoretical maximum.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: [mmol/l.min]
Arm/Group | Placebo | Melatonin
Number analyzed (Participants) | 21 | 20
[mmol/l.min] | 322.6 (24.7) [296.5 to 350.9] | 329.4 (12.7) [302.9 to 358.2]

ADVERSE EVENTS:
Time Frame: From admission to the in-laboratory until the discharge from the laboratory, up to 5 days
Description: Adverse events were reported with both interventions combined. This is because the adverse events happened either before any intervention started or after both ended, it is hard to attribute the events to one specific intervention.
Groups:
- All Intervention Combined: Placebo or Melatonin oral administration on Day 2 or Day 4 of their in-laboratory stay (order randomized)
Arm/Group | All Intervention Combined
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 2/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Intervention Combined (N=23)
Nausea (General disorders) | 1 — Participant felt nausea when consuming test breakfast
Failed attempts to place IV lines (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT02642640/Prot_SAP_000.pdf